CLINICAL TRIAL: NCT02920606
Title: Pulpotomy as a Permanent Treatment of Irreversible Pulpitis on Mature Molar Teeth - a Pilot Study
Brief Title: Pulpotomy as a Treatment of Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pulpotomie-1
Record Dates: First submitted 2016-05-30; First posted 2016-09-30 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Irreversible Pulpitis
Keywords: pulpotomy; pulpitis; mature tooth; tricalcium silicate
MeSH Terms: conditions — Pulpitis | interventions — Pulpotomy; Endodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endodontic treatment (Active Comparator): The patient will benefit from a conventional treatment : a root canal treatment.
  The root canal treatment consists of removing the pulp tissue from all the canals, disinfecting the root canal system with sodium hypochlorite and filling the root with a root canal sealer and gutta percha.
  Interventions: Procedure: Endodontic treatment
- Pulpotomy (Experimental): The patient will benefit from an experimental treatment : a pulpotomy. The pulpotomy aims at removing the coronal part of the pulp (the pulp present in the pulp chamber) and filling the pulp chamber with a bioactive material.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy
  Arms: Pulpotomy
Procedure: Endodontic treatment
  Arms: Endodontic treatment

SUMMARY:
The procedure currently recommended for the treatment of irreversible pulpitis is the endodontic treatment, i.e. the complete elimination of the pulp, disinfection and obturation of the whole root canal system. The emergency procedure consists of a pulpotomy, followed at an ulterior appointment by the root canal treatment. The purpose of the present pilot study is to evaluate the feasibility of performing the pulpotomy as a permanent treatment in mature molars. If hemostasis can be achieved after removing the coronal part of the pulp, a tricalcium silicate cement will be directly applied on the remaining pulp at the root canal entrances. A short-term follow-up will be performed at one week by evaluating the pain relief of the patient. Long-term success will then be evaluated every year by verifying the absence of periapical radiolucency on the x-ray as well as the absence of clinical symptoms and signs. A standard root canal procedure will serve as control. During the pulpotomy treatment, blood sample with microcapillary will be performed. We will analyze a ratio of pro-inflammatory and anti-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Not pregnant women
* At least one permanent molar in irreversible pulpitis
* Adult patient
* Mentally competent

Exclusion Criteria:

* Periapical radiolucency
* Periodontical probing
* Root fracture
* Sinus tract
* Swelling or mobility
* External or/and internal resorption
* Open apicies
* A non restorable tooth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the success rate (%) at 1 year | Follow up at 1 year for all patients included in the study
  to evaluate the treatment success defined as the absence of clinical symptoms (pain, sinus tract..) and the absence of radiological symptoms (periapical radiolucency), in order to point the non-inferiority of the pulpotomy compared with the conventional treatment

SECONDARY OUTCOMES:
Evaluation of the correlation between pro/anti-inflammatory cytokines and the success of pulpotomy | Follow up at 1 year for all patients included in the study
  During the pulpotomy treatment, blood samples with microcapillaries will be performed. We will analyze a ratio of pro-inflammatory and anti-inflammatory cytokines.

OTHER OUTCOMES:
Evaluation of the success rate (%) up to 4 years | Follow up at 4 years for all patients included in the test group
  to evaluate the treatment success defined as the absence of clinical symptoms (pain, sinus tract..) and the absence of radiological symptoms (periapical radiolucency), in order to point the non-inferiority of the pulpotomy compared with the conventional treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julian G Leprince, Professor, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No